CLINICAL TRIAL: NCT06953596
Title: Transcranial Magnetic Stimulation to Treat Prolonged Grief Disorder: A Single-centre, Single-arm, Open-label Phase I/II Proof-of-concept and Feasibility Clinical Trial
Brief Title: Transcranial Magnetic Stimulation to Treat Prolonged Grief Disorder
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bruyère Health Research Institute. (Other)
Responsible Party: Principal Investigator, James Downar, Head, Division of Palliative Care, University of Ottawa, Bruyère Health Research Institute.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23732836368
Record Dates: First submitted 2025-04-22; First posted 2025-05-01 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Prolonged Grief Disorder; Complicated Grief
Keywords: Neuromodulation; Repetitive Transcranial Magnetic Stimulation; Bereavement; Proof-of-Concept; Feasibility; Intermittent Theta Burst Stimulation (iTBS)
MeSH Terms: conditions — Prolonged Grief Disorder | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: Single-centre, single-arm, open-label phase I/II proof-of-concept and feasibility clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- rTMS Intervention (Experimental)
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation (rTMS)

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation (rTMS) — Eight rTMS sessions will be administer per day at 60-minute intervals for 5 consecutive days.
  Each rTMS session will consist of 600 pulses of theta-burst stimulation (iTBS), a pattern of 3 TMS pulses every 200 milliseconds for 2 seconds (i.e., 3 x 50 Hz bursts repeated at 5 Hz) for 3 minutes at 100% of resting motor threshold. The left dorsomedial prefrontal cortex (DMPFC) will be targeted via the Fz EEG site (30% of the nasion-inion distance posteriorly along the nasion-inion line).

SUMMARY:
Grief is a normal response after the death of a loved one. With time, the grief response decreases and people learn to cope with their loss. However, for some, the response becomes more intense and distressing. This is called prolonged grief disorder (PGD). People with PGD experience emotional pain and a deep longing for their loved one. PGD normally occurs <10% of people after a loss, but it has become more common since the COVID-19 pandemic (~30%). If left untreated, PGD leads to poor quality of life and increased risk of death. Treatment options such as medication and therapy are available; however, they can cause negative side effects and take a long time to work. To help individuals with PGD, we need treatments that work well and quickly.

Repetitive transcranial magnetic stimulation (rTMS) is a safe, non-invasive treatment that delivers magnetic pulses to brain areas responsible for mood. rTMS has been approved in Canada to treat mood disorders. There is research to show that rTMS is safe and well-tolerated, and that works well in treating Post-Traumatic Stress Disorder (PTSD), a condition with similar symptoms to PGD. To determine whether rTMS is effective for treating PGD, we first need to determine if rTMS as a treatment for PGD is safe and feasible among grieving individuals.

DETAILED DESCRIPTION:
Prolonged Grief Disorder (PGD) is an important challenge among bereaved individuals. While the grief response following loss is typically acute, with symptoms diminishing over time, it can sometimes lead to prolonged grief disorder (PGD). PGD is characterized by persistent longing and preoccupation with the decedent, emotional pain, as well as cognitive and functional impairment that persists for more than 6 months after a loss. Prevalence rates for PGD vary; systematic reviews show pooled prevalence rates of 10% after death due to natural causes, but rising as high as 49% after death due to sudden or violent causes (e.g., suicide, homicide, mass casualty event). We found that the incidence of PGD in the COVID-19 pandemic rose to ~30% of bereaved family members, regardless of the cause of death (COVID-19 or other illness), and that the prevalence remained unchanged more than 18 months post-loss. PGD is also more common among women, people with severe pre-loss grief or depressive symptoms, those who have lost a child, and those with structural vulnerability (e.g. lower education level and income). Recently, PGD was included as a diagnostic entity in the International Classification of Diseases (ICD), and the Diagnostic and Statistical Manual of Mental Disorders (DSM).

PGD is associated with serious physical and mental health problems, including increased incidence of cardiovascular events, sleep disturbances, substance abuse, and suicidal ideation, resulting in poor overall quality of life and increased risk of mortality. Alongside the physical and psychological symptoms of bereavement, there is a concomitant increase in healthcare utilization, contributing to increased healthcare expenditure. PGD has been associated with increased emergency department visits, general hospital admissions, psychiatric hospitalizations, general practitioner, psychiatrist, and psychologist visits, as well as use of medications such as antidepressants and anxiolytics. Studies have shown that bereaved individuals have increased healthcare expenditures compared to non-bereaved controls, and widowed individuals spend 40% more on healthcare during the first 2-years post-death compared with pre-death expenditures. Moreover, bereaved individuals are less economically productive, particularly when they have PGD. In response to the accumulating evidence showing the wide-reaching consequences of PGD, several organizations (e.g., Canadian Grief Alliance, Canadian Virtual Hospice), are calling for the development and implementation of a national grief strategy to address this "hidden and urgent public health crisis."

Existing treatment options for PGD are limited. Pharmacotherapies such as antidepressants (e.g., tricyclic antidepressants, selective serotonin reuptake inhibitors) are often prescribed for PGD, though their efficacy for grief-related symptoms is minimal, and time to effect and side effects (e.g., headaches, dry mouth, insomnia, flashbacks, palpitations) are barriers to uptake. Psychotherapy (including Complicated Grief Therapy) has shown moderate effectiveness in symptom reduction in a small number of trials, but issues with homogenous (e.g., primarily Western countries) and small samples and variable inclusion criteria raise questions about the generalizability of the evidence. Additionally, psychotherapy is resource-intensive and time-consuming with delayed effectiveness. There is an acute need for feasible, effective, and scalable treatment options to respond to PGD.

Repetitive Transcranial Magnetic Stimulation (rTMS) may be a feasible and efficacious treatment for PGD. rTMS is a safe, tolerable, and non-invasive brain stimulation technique approved by Health Canada in 2002 for the treatment of major depression, post-traumatic stress disorder (PTSD), and other mood and anxiety disorders. Using an inductor coil placed against the scalp, rTMS employs powerful, focused magnetic pulses to induce an electrical current that depolarizes the underlying neuronal tissue and causes action potentials which, depending on the stimulation parameters (high-frequency vs. low-frequency), increase or decrease cortical excitability. When administered repetitively, TMS can cause long-term neuromodulation and subsequent therapeutic benefit.

rTMS is effective for treating post-traumatic stress disorder (PTSD). To date, over 15 studies (10 RCTs) have demonstrated safety, tolerability, efficacy, and durability for treating PTSD with high- and low-frequency rTMS stimulation at different sites (e.g., right dorsolateral prefrontal cortex (DLPFC), left DLPFC, and medial prefrontal cortex).Notably, one open-label case series reported >50% improvement in PTSD symptoms in 57% of patients following rTMS to the dorsomedial prefrontal cortex. However, rTMS has never been evaluated for the treatment of PGD. Clinically, experiences associated with PGD (i.e., trauma associated with the dying and grief experience) and its symptoms are similar to PTSD, with several overlapping characteristics (e.g., intrusive thoughts or images, avoidance, emotional numbness), raising the question of whether rTMS may be efficacious for treating PGD too.

Objective:

To determine if accelerated rTMS is a safe and feasible treatment for PGD among bereaved individuals. The secondary objective is to examine the preliminary efficacy of accelerated rTMS for treatment of PGD.

Sample Size:

As the main objective of this study is to demonstrate safety and feasibility, no formal sample size calculation was performed. The goal of this study is to provide estimates, along with margins of error, of the enrollment rate and efficacy outcomes to inform a subsequent sham-controlled clinical trial.

Statistical Analysis:

Analysis of safety and feasibility outcomes will be descriptive, with point estimates and 95% confidence intervals. The efficacy analysis will follow an intent-to-treat approach. We will compare the proportion of participants with a minimal clinically important difference in secondary efficacy outcomes at 2-week follow-up.

Details of Eligibility, Intervention Protocol, and Outcome Measures are provided elsewhere.

ELIGIBILITY:
Inclusion Criteria:

1. Bereaved individuals >/= 18 years of age
2. Score >25 on the Inventory of Complicated Grief
3. Must have a primary care physician
4. Ability to understand and communicate in English
5. Ability to provide first-person informed consent

Exclusion Criteria:

1. Current or previously diagnosed seizure disorder
2. Documented brain lesions
3. Contraindications to TMS (i.e., metallic skull plates, clips, stimulators, pacemakers)
4. Current substance abuse disorder (e.g., schizophrenia)
5. Pregnancy or lactation, or trying to conceive
6. Advanced, incurable illness with an expected prognosis of <3 months - bereaved family members are known to be at elevated risk of death from medical illness, but if death is expected in the near future, it would be difficult to justify using an entire week of their limited time for an unproven therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Recruitment Rate | Through study completion, up to 9 months
  Number of individuals recruited divided by the recruitment period
Enrollment Rate | Through study completion, up to 9 months
  Number of individuals enrolled divided by the number of individuals approached
Intervention Completion Rate | Through study completion, up to 10 months
  Number of participants who complete the intervention divided by the number of participants enrolled
Withdrawal Rate | Through study completion, up to 16 months
  Number of participants who withdrew divided by the number of participants enrolled
Follow-up Completion Rate | Through study completion, up to 16 months
  Number of participants who complete follow-up divided by the number of participants enrolled
Number of Participants with Adverse Events | Through intervention completion, up to 1 week
  Proportion of participants who experience an adverse event

SECONDARY OUTCOMES:
Prolonged Grief Disorder - Global Impression of Change | Day 5 (last day of intervention), 2-week follow-up, 4-week follow-up, and monthly thereafter for up to 6 months
  Measured using the Patient Global Impression of Change (PGIC) scale (score 1-7 on one item; higher scores indicate greater positive change)
Change in Prolonged Grief | Baseline, day 5 (last day of intervention), 2-week follow-up, 4-week follow-up, and monthly thereafter for up to 6 months
  Measured using the Inventory of Complicated Grief (ICG) (score 0-4 on each item; score of 26 or less or a score reduction of greater than or equal to 4 indicates therapeutic benefits)
Prolonged Grief - Change in Post-Traumatic Stress | Baseline, day 5 (last day of intervention), 2-week follow-up, 4-week follow-up, and monthly thereafter for up to 6 months
  Measured using the Impact of Event Scale-Revised (IES-R) (score 0-4 on each item; score reduction of 4 indicates therapeutic benefit; score greater than 33 will be considered positive for PTSD)
Prolonged Grief - Change in Depression | Baseline, day 5 (last day of intervention), 2-week follow-up, 4-week follow-up, and monthly thereafter for up to 6 months
  Measured using the Hamilton Depression Rating Scale (HDRS) (score 0-4 on each item; score reduction of 2 from baseline indicates therapeutic benefit)
Prolonged Grief - Change in Work and Social Functioning | Baseline, day 5 (last day of intervention), 2-week follow-up, 4-week follow-up, and monthly thereafter for up to 6 months
  Measured using the Work and Social Adjustment Scale (WSAS) (score of 0-8 on each item; point difference of greater than or equal to 8 indicates therapeutic benefit)

CONTACTS AND LOCATIONS:
Locations (1):
- Bruyere Health, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Prigerson HG, Bierhals AJ, Kasl SV, Reynolds CF 3rd, Shear MK, Day N, Beery LC, Newsom JT, Jacobs S. Traumatic grief as a risk factor for mental and physical morbidity. Am J Psychiatry. 1997 May;154(5):616-23. doi: 10.1176/ajp.154.5.616. PMID 9137115
- [Background] Szuhany KL, Malgaroli M, Miron CD, Simon NM. Prolonged Grief Disorder: Course, Diagnosis, Assessment, and Treatment. Focus (Am Psychiatr Publ). 2021 Jun;19(2):161-172. doi: 10.1176/appi.focus.20200052. Epub 2021 Jun 17. PMID 34690579
- [Background] Buur C, Zachariae R, Komischke-Konnerup KB, Marello MM, Schierff LH, O'Connor M. Risk factors for prolonged grief symptoms: A systematic review and meta-analysis. Clin Psychol Rev. 2024 Feb;107:102375. doi: 10.1016/j.cpr.2023.102375. Epub 2023 Dec 29. PMID 38181586
- [Background] Lapenskie J, Anderson K, Lawlor PG, Kabir M, Noel C, Heidinger B, Parsons HA, Cohen L, Gratton V, Besserer E, Adeli S, Murphy R, Warmels G, Bruni A, Bhimji K, Dyason C, Enright P, Desjardins I, Wooller K, Arsenault-Mehta K, Webber C, Bedard D, Iyengar A, Bush SH, Isenberg SR, Tanuseputro P, Vanderspank-Wright B, Downar J. Long-term bereavement outcomes in family members of those who died in acute care hospitals before and during the first wave of COVID-19: A cohort study. Palliat Med. 2024 Feb;38(2):264-271. doi: 10.1177/02692163231223394. Epub 2024 Jan 16. PMID 38229211
- [Background] Downar J, Parsons HA, Cohen L, Besserer E, Adeli S, Gratton V, Murphy R, Warmels G, Bruni A, Bhimji K, Dyason C, Enright P, Desjardins I, Wooller K, Kabir M, Noel C, Heidinger B, Anderson K, Arsenault-Mehta K, Lapenskie J, Webber C, Bedard D, Iyengar A, Bush SH, Isenberg SR, Tanuseputro P, Vanderspank-Wright B, Lawlor P. Bereavement outcomes in family members of those who died in acute care hospitals before and during the first wave of COVID-19: A cohort study. Palliat Med. 2022 Sep;36(8):1305-1312. doi: 10.1177/02692163221109711. Epub 2022 Jul 4. PMID 35786109
- [Background] Djelantik AAAMJ, Smid GE, Mroz A, Kleber RJ, Boelen PA. The prevalence of prolonged grief disorder in bereaved individuals following unnatural losses: Systematic review and meta regression analysis. J Affect Disord. 2020 Mar 15;265:146-156. doi: 10.1016/j.jad.2020.01.034. Epub 2020 Jan 13. PMID 32090736
- [Background] Lundorff M, Holmgren H, Zachariae R, Farver-Vestergaard I, O'Connor M. Prevalence of prolonged grief disorder in adult bereavement: A systematic review and meta-analysis. J Affect Disord. 2017 Apr 1;212:138-149. doi: 10.1016/j.jad.2017.01.030. Epub 2017 Jan 23. PMID 28167398
- [Background] Kentish-Barnes N, Prigerson HG. Is this bereaved relative at risk of prolonged grief? Intensive Care Med. 2016 Aug;42(8):1279-81. doi: 10.1007/s00134-015-4182-6. Epub 2015 Dec 23. No abstract available. PMID 26699916
- [Background] Lenferink LIM, van den Munckhof MJA, de Keijser J, Boelen PA. DSM-5-TR prolonged grief disorder and DSM-5 posttraumatic stress disorder are related, yet distinct: confirmatory factor analyses in traumatically bereaved people. Eur J Psychotraumatol. 2021 Dec 9;12(1):1-14. doi: 10.1080/20008198.2021.2000131. eCollection 2021. PMID 34912501
- [Background] Shear MK, Simon N, Wall M, Zisook S, Neimeyer R, Duan N, Reynolds C, Lebowitz B, Sung S, Ghesquiere A, Gorscak B, Clayton P, Ito M, Nakajima S, Konishi T, Melhem N, Meert K, Schiff M, O'Connor MF, First M, Sareen J, Bolton J, Skritskaya N, Mancini AD, Keshaviah A. Complicated grief and related bereavement issues for DSM-5. Depress Anxiety. 2011 Feb;28(2):103-17. doi: 10.1002/da.20780. PMID 21284063
- [Background] Tang S, Xiang Z. Who suffered most after deaths due to COVID-19? Prevalence and correlates of prolonged grief disorder in COVID-19 related bereaved adults. Global Health. 2021 Feb 11;17(1):19. doi: 10.1186/s12992-021-00669-5. PMID 33573673
- [Background] Prigerson HG, Kakarala S, Gang J, Maciejewski PK. History and Status of Prolonged Grief Disorder as a Psychiatric Diagnosis. Annu Rev Clin Psychol. 2021 May 7;17:109-126. doi: 10.1146/annurev-clinpsy-081219-093600. Epub 2021 Feb 1. PMID 33524263